CLINICAL TRIAL: NCT04884919
Title: Develop the First Aid Medical Supplies for Hemostasis and Bacteriostasis With Clinical Trial
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Tri-Service General Hospital (Other)
Responsible Party: Principal Investigator, Hsu Sheng-Der, Attending Physician, Tri-Service General Hospital
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Chitosan-Microbiome
Record Dates: First submitted 2021-05-02; First posted 2021-05-13 (Actual); Last update posted 2021-05-13 (Actual); Status verified 2021-05

CONDITIONS: Cesarean Section

STUDY DESIGN:
Intervention Model Description: Each of the participants is treated with 2 different treatments on different areas of the same wound at the same time.
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Regular Gauze Treatment (Placebo Comparator): Participants who undergo a cesarean section are first dissected in about 5 cm length and 2 cm width and receive a regular gauze made of traditional cotton yarn. The regular gauze is applied on the half side of the wound.
  Interventions: Device: Regular Gauze
- Chitosan Dressing Treatment (Experimental): Participants who undergo a cesarean section are first dissected in about 5 cm length and 2 cm width and receive a chitosan dressing made of chitosan material. The chitosan dressing is applied on another half side of the wound.
  Interventions: Device: Chitosan Dressing

INTERVENTIONS:
Device: Regular Gauze — Regular gauze
  Arms: Regular Gauze Treatment
Device: Chitosan Dressing — Dressing made of chitosan material
  Arms: Chitosan Dressing Treatment

SUMMARY:
The current development of hemostatic and open wound infection care strategies will focus on enhancing the efficiency of hemostasis for internal bleeding, relieving pain, avoiding wound infection, and promoting wound healing. As the social environment changes, the demand for hemostatic techniques and wound healing is increasing. Thus, hemostatic techniques are needed to be integrated with functional functions for usual trauma care, and the wound care strategies that can inhibit and reduce infection while helping to facilitate wound healing are needed to be developed to ensure the safety of human life. Therefore, this trial aims to develop new biofiber hemostatic dressings for hemostasis and open wound care. The comparisons of hemostatic and antibacterial effects, hemostatic time, wound infection status, wound bacteria count, and wound adhesion situation obtained from this clinical trial are expected able to establish a better rapid hemostatic strategy and wound infection care strategy.

DETAILED DESCRIPTION:
This trial is performed when the subjects undergoing a cesarean section at Tri-Service General Hospital, Taipei, Taiwan (R.O.C). After disinfection of the surgical wound, regular gauze and chitosan dressings are directly and simultaneously placed over the disinfected wound with finger pressure for 3 min, immediately after the dissection. The regular gauze dressing is placed on half side of the surgical wound, while the chitosan dressing is placed on another half side of the wound. After 3 min, the pressure is stopped and the doctors will photograph and observe both dressings whether the bleeding has stopped. If the bleeding on the surface of the wound has stopped after 20 s, the bleeding is considered to have stopped and the wound is then treated according to the scheduled surgical procedure. If the bleeding has not stopped, finger pressure to stop bleeding will be given for 5 min. Then, after 5 minutes, the pressure is stopped and the bleeding condition is observed. If the bleeding has stopped after 20 s, the bleeding of the wound is judged to have stopped and the subsequent surgery will be performed. However, if it still bleeds, both dressings will be replaced and do the same for another 5 min. (Note) Depending on the physiological parameters of each patient, the decision can be determined by the physician; if bleeding or hematoma occurs, the patient will be treated according to hospital procedure until the symptoms are relieved, and evaluate whether the test should be stopped.

The postoperative wound will be dressed with regular gauze and chitosan dressings and the wound condition will be recorded on day 0 of the trial. The dressing is daily changed by replacing regular gauze and chitosan dressings and by performing wound care. The test of the dressing sample will be taken for bacterial analysis. If there are symptoms of infection after 14 days of this test, the wound will be treated in accordance with the clinical routine wound treatment. (Note) If the wound condition shows serious infection during the dressing change process, the treatment should be carried out according to the clinical routine treatment method, and it is determined and evaluated whether to stop the test. (Note) If the patient's psychological stress is affected during the trial, the physician will explain and determine whether the trial must be stopped.

ELIGIBILITY:
Inclusion Criteria:

* The subject is aged between 20 and 80 years old.
* Patients who need a cesarean section.
* The expected size of the wound is about 5 cm or more in length and 2 cm or more in width.

Exclusion Criteria:

* Patients with a history of allergy to chitin components such as shrimp and crab.
* Patients with blood clotting disorders.
* Vulnerable groups.
* Patients with unstable signs of life.

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2019-05-10 (Actual); Primary Completion 2021-12-31 (Estimated); Study Completion 2021-12-31 (Estimated)

PRIMARY OUTCOMES:
Hemoglobin Assay | 3 up to 13 minutes
  After 3, 5, and additional 5 minutes, consecutively depending on the patients' conditions, the use of regular gauze and chitosan dressings to compress the abdominal surgical wounds are incubated in jars containing 0.9% (w/v) saline solution for 1, 3, 5, and 10 minutes, respectively. 1 mL solution of the dressing incubation is collected and evaluated using a hemoglobin standard (H7379, Sigma-Aldrich; Merck KGaA, Darmstadt, Germany). The hemoglobin concentration is measured by examining the optical density at 540 nm wavelength.
Adenosine Triphosphate (ATP) Assay | Up to 8 days
  This assay is performed to evaluate and compare antimicrobial properties of both dressings. Adenosine triphosphate (ATP) bioluminescence assay expressed in Relative Fluorescence Units (RFU) is used to measure the number of bacteria by using ATP luminometer (LuciPac Pen PD 30, Kikkoman Biochemifa Co., Tokyo, Japan).
Phylogenetic of Microbial Community | Up to 3 days
  Wound-contacted dressings of patients are collected on day 1 and day 3 postoperation and kept at 4°C within an hour processed for genomic DNA isolation using DNeasy Blood & Tissue kit (QIAGEN, Germany). Amplification of 16S-rRNA-genes of distinct regions V3-V4 is conducted using specific primer 16S V3+V4: 314F-806R with the barcode. Phusion® High-Fidelity PCR Master Mix (New England Biolabs) is then used for all PCR reactions. Subsequently, 300bp paired-end raw reads are implemented for amplicon sequencing. Finally, the entire paired-end reads are incorporated using FLASH v.1.2.7.
Heat Map Analysis | Up to 6 days
  The heat map is analyzed using an R package to acquire the distribution of bacteria population in wound-contacted dressings. This analysis results the distribution of heat produced by bacteria population that is scaled from -1 to 1 indicating the abundance of each genus of bacteria from the lowest temperature to the highest temperature.
Partial Least Squares Discriminant Analysis (PLS-DA) | Up to 6 days
  PLS-DA is analyzed using PLS toolbox (Eigenvector Research Incorporated Wenatchee, WA, USA) for Matlab® R2009b software (Mathworks Inc., Natick MA, USA) to get the discriminant of bacterial community between the wound-contacted dressing.
UpSet Plot | Up to 6 days
  The UpSet plot of Bacteria Operational Taxonomy Units is produced in R using UpSetR. This results intersection sizes of bacteria among the experiment groups.
Statistical Analysis | Up to 8 days
  Statistical calculations are performed using SPSS software version 21 (SPSS, Chicago, IL, USA) and written in the form of mean ± standard error of the mean. Data means are compared by one-way or two-way analysis of variance (ANOVA) among two or more than two groups for statistical comparison. The significance level is set at p < 0.05.

CONTACTS AND LOCATIONS:
Locations (1):
- National Defense of Medical Center, Tri-Service General Hospital, Taipei, Taiwan

REFERENCES:
- [Background] Kang X, Liu G, Liu Y, Xu Q, Zhang M, Fang M. Transcriptome profile at different physiological stages reveals potential mode for curly fleece in Chinese tan sheep. PLoS One. 2013 Aug 26;8(8):e71763. doi: 10.1371/journal.pone.0071763. eCollection 2013. PMID 23990983
- [Background] Chen B, Gao LL, Pan Q. Woody forages effect the intestinal bacteria diversity of golden pompano Trachinotus ovatus. AMB Express. 2018 Feb 27;8(1):29. doi: 10.1186/s13568-018-0550-2. PMID 29484505
- [Background] Vijayalakshmi S, Adeyemi DE, Choi IY, Sultan G, Madar IH, Park MK. Comprehensive in silico analysis of lactic acid bacteria for the selection of desirable probiotics. LWT. 2020; 130:109617.
- [Background] Akanny, E, Bonhommé, A, Commun, C, et al. Surface-enhanced Raman spectroscopy using uncoated gold nanoparticles for bacteria discrimination. J Raman Spectrosc. 2020; 51: 619- 629.
- [Background] Ramadan Z, Jacobs D, Grigorov M, Kochhar S. Metabolic profiling using principal component analysis, discriminant partial least squares, and genetic algorithms. Talanta. 2006 Feb 28;68(5):1683-91. doi: 10.1016/j.talanta.2005.08.042. Epub 2005 Sep 19. PMID 18970515
- [Background] Ruparell A, Inui T, Staunton R, Wallis C, Deusch O, Holcombe LJ. The canine oral microbiome: variation in bacterial populations across different niches. BMC Microbiol. 2020 Feb 28;20(1):42. doi: 10.1186/s12866-020-1704-3. PMID 32111160